CLINICAL TRIAL: NCT02010775
Title: BOTOX® Treatment of Masseter Muscle Hypertrophy
Brief Title: Botulinum Toxin Type A (BOTOX®) Treatment of Masseter Muscle Hypertrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191622-130
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-02

CONDITIONS: Masseter Muscle Hypertrophy
MeSH Terms: conditions — Masticatory Muscles, Hypertrophy of | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- BOTOX® 24U (Active Comparator): Botulinum Toxin Type A (BOTOX®) 24U total dose administered intramuscularly to the bilateral masseter muscles on Day 1 and retreatment at Day 180 if applicable.
  Interventions: Biological: botulinum toxin Type A
- BOTOX® 48U (Active Comparator): Botulinum Toxin Type A (BOTOX®) 48U total dose administered intramuscularly to the bilateral masseter muscles on Day 1 and retreatment at Day 180 if applicable.
  Interventions: Biological: botulinum toxin Type A
- BOTOX® 72U (Active Comparator): Botulinum Toxin Type A (BOTOX®) 72U total dose administered intramuscularly to the bilateral masseter muscles on Day 1 and retreatment at Day 180 if applicable.
  Interventions: Biological: botulinum toxin Type A
- BOTOX® 96U (Active Comparator): Botulinum Toxin Type A (BOTOX®) 96U total dose administered intramuscularly to the bilateral masseter muscles on Day 1 and retreatment at Day 180 if applicable.
  Interventions: Biological: botulinum toxin Type A
- Placebo (Placebo Comparator): Placebo (Normal saline) administered intramuscularly to the bilateral masseter muscles on Day 1 and retreatment at Day 180 if applicable.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Biological: botulinum toxin Type A — Botulinum toxin Type A (BOTOX®) administered intramuscularly to the bilateral masseter muscles on Day 1 and retreatment at Day 180 if applicable.
  Other Names: BOTOX®; onabotulinumtoxinA
  Arms: BOTOX® 24U; BOTOX® 48U; BOTOX® 72U; BOTOX® 96U
Drug: Normal saline — Normal saline (placebo) administered intramuscularly to the bilateral masseter muscles.
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of a range of doses of botulinum toxin Type A (BOTOX®) for the treatment of patients with bilateral Masseter Muscle Hypertrophy (MMH).

ELIGIBILITY:
Inclusion Criteria:

-Participants with Masseter Muscle Hypertrophy

Exclusion Criteria:

* Diagnosis of Myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function
* Prior botulinum toxin treatment of any serotype to the masseter muscle or lower face
* History of dental or surgical procedure for lower facial shaping or masseter muscle reduction
* History of or current temporomandibular joint disorder (TMJD)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 187 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beta Bowen, Study Director — Allergan
Locations (14):
- Australia (4):
  - Shape Clinic, Darlinghurst, New South Wales
  - Central Sydney Dermatology, Sydney, New South Wales
  - Esteem Beauty & Day Spa, Main Beach, Queensland
  - The Rose Medical & Aesthetic Centre, North Fremantle, Western Australia
- Canada (6):
  - Dr. Jean Carruthers Cosmetic Surgery, Inc., Vancouver, British Columbia
  - Dr. Shannon Humphrey Inc., Vancouver, British Columbia
  - Project Skin MD, Vancouver, British Columbia
  - Pacific Dermaesthetics, Vancouver, British Columbia
  - Bertucci MedSpa, Woodbridge, Ontario
  - Arthur Swift Research Inc., Montreal, Quebec
- Taiwan (4):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Taipei Chang Gung Memorial Hospital of CGMF, Taipei
  - Tri-Service General Hospital, Taipei

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BOTOX® 96U | BOTOX® 72U | BOTOX® 48U | BOTOX® 24U | Placebo
Started | 38 | 38 | 37 | 37 | 37
Completed | 33 | 35 | 34 | 34 | 31
Not Completed | 5 | 3 | 3 | 3 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 1 | 1
Not completed — Personal Reasons | 3 | 3 | 1 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population included all randomized participants who received at least 1 injection of study treatment and had at least 1 follow-up visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | BOTOX® 96U | BOTOX® 72U | BOTOX® 48U | BOTOX® 24U | Placebo | Total
Number analyzed (Participants) | 38 | 38 | 37 | 37 | 37 | 187
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.3 (9.10) | 34.9 (8.35) | 37.2 (7.69) | 34.0 (9.08) | 35.4 (8.08) | 35.4 (8.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 31 | 32 | 32 | 153
  Male | 8 | 10 | 6 | 5 | 5 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 7 | 7 | 7 | 5 | 10 | 36
  Asian | 30 | 30 | 30 | 32 | 27 | 149
  Hispanic | 0 | 1 | 0 | 0 | 0 | 1
  Other Race | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lower Facial Volume Using VECTRA 3D Images
Description: Lower facial volume was calculated from 3-dimensional (3D) images captured with the VECTRA M3 3D Stereophotogrammetry imaging system and was analyzed using computer assisted systems and predetermined facial landmarks. The difference in volume was measured between the select region of the baseline surface 3D model and the select region of the posttreatment surface 3D model. A negative change from Baseline (decrease in volume) indicates improvement.
Time Frame: Baseline (Day 1) to Day 90 of Treatment Cycle 1
Population: Participants from the mITT population, all randomized participants who received at least 1 injection of study treatment and had at least 1 follow-up visit, with data available for analysis at Day 90. Change in lower facial volume was quantified in cm^3 using image subtraction techniques; as the Baseline is an image, no Baseline data are reported.
Measure: Least Squares Mean (Full Range); unit: cubic centimeter (cm^3)
Arm/Group | BOTOX® 96U | BOTOX® 72U | BOTOX® 48U | BOTOX® 24U | Placebo
Number analyzed (Participants) | 38 | 38 | 36 | 36 | 37
cubic centimeter (cm^3) | -8.20 [-15.6 to -1.4] | -7.41 [-16.5 to -0.8] | -6.84 [-17.4 to 1.6] | -4.40 [-13.2 to 2.0] | -0.52 [-6.7 to 9.0]
Statistical Analysis 1: Comparison: BOTOX® 24U vs Placebo; Test type: Other; p < 0.001, ANOVA; ANOVA model with treatment, and baseline MMPS grade as factors; Least Squares Mean (LS) Mean Difference = -3.88, 95% CI 2-sided [-5.58 to -2.19]
Statistical Analysis 2: Comparison: BOTOX® 48U vs Placebo; Test type: Other; p < 0.001, ANOVA; ANOVA model with treatment, and baseline MMPS grade as factors; LS Mean Difference = -6.32, 95% CI 2-sided [-8.02 to -4.62]
Statistical Analysis 3: Comparison: BOTOX® 72U vs Placebo; Test type: Other; p < 0.001, ANOVA; ANOVA model with treatment, and baseline MMPS grade as factors; LS Mean Difference = -6.89, 95% CI 2-sided [-8.56 to -5.22]
Statistical Analysis 4: Comparison: BOTOX® 96U vs Placebo; Test type: Other; p < 0.001, ANOVA; ANOVA model with treatment, and baseline MMPS grade as factors; LS Mean Difference = -7.68, 95% CI 2-sided [-9.35 to -6.00]

2. Secondary Outcome: Percentage of Participants Who Achieved a Masseter Muscle Prominence Scale (MMPS) Grade ≤ 3 as Assessed by the Investigator
Description: The investigator used visual inspection and palpation to grade the prominence of the participant's masseter muscle on the left and right sides of the face using the MMPS where: 1=minimal prominence (best), 2=mild prominence, 3=moderate prominence, 4=marked prominence, 5=very marked prominence (worst). The percentage of participants with grade 3 or less is reported.
Time Frame: Day 90 of Treatment Cycle 1
Population: Participants from the mITT population, all randomized participants who received at least 1 injection of study treatment and had at least 1 follow-up visit, with data available for analysis at Day 90. Missing data was imputed using last observation carried forward.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BOTOX® 96U | BOTOX® 72U | BOTOX® 48U | BOTOX® 24U | Placebo
Number analyzed (Participants) | 38 | 38 | 36 | 36 | 37
Percentage of participants | 89.5 [75.2 to 97.1] | 89.5 [75.2 to 97.1] | 83.3 [67.2 to 93.6] | 66.7 [49.0 to 81.4] | 35.1 [20.2 to 52.5]
Statistical Analysis 1: Comparison: BOTOX® 24U vs Placebo; Test type: Other; p = 0.008, Cochran-Mantel-Haenszel; P-values for between-treatment comparisons were determined using Cochran-Mantel-Haenszel (CMH) tests stratified by baseline MMPS; Percentage Difference = 31.5, 95% CI 2-sided [9.8 to 53.3]
Statistical Analysis 2: Comparison: BOTOX® 48U vs Placebo; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; P-values for between-treatment comparisons were determined using CMH tests stratified by baseline MMPS; Percentage Difference = 48.2, 95% CI 2-sided [28.6 to 67.8]
Statistical Analysis 3: Comparison: BOTOX® 72U vs Placebo; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; P-values for between-treatment comparisons were determined using CMH tests stratified by baseline MMPS; Percentage Difference = 54.3, 95% CI 2-sided [36.1 to 72.6]
Statistical Analysis 4: Comparison: BOTOX® 96U vs Placebo; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; P-values for between-treatment comparisons were determined using CMH tests stratified by baseline MMPS; Percentage Difference = 54.3, 95% CI 2-sided [36.1 to 72.6]

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) to the end of study (Month 12)
Description: Safety Population, all treated participants based on the treatment received, was used to determine the number of participants at risk for Serious Adverse Events and Adverse Events.
Arm/Group | BOTOX® 96U | BOTOX® 72U | BOTOX® 48U | BOTOX® 24U | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38 | 0/37 | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 1/38 | 0/38 | 0/37 | 2/37 | 3/37
Other Adverse Events (participants affected / at risk) | 13/38 | 10/38 | 12/37 | 16/37 | 10/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | BOTOX® 96U (N=38) | BOTOX® 72U (N=38) | BOTOX® 48U (N=37) | BOTOX® 24U (N=37) | Placebo (N=37)
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Uterine leiomyomax (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/30 | 0/28 | 0/31 | 0/32 | 1/32 — For this gender-specific preferred term, percentages were calculated based on gender-specific denominators for females.
Abortion induced (Surgical and medical procedures) | 0/30 | 0/28 | 0/31 | 1/32 | 0/32 — For this gender-specific preferred term, percentages were calculated based on gender-specific denominators for females.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® 96U (N=38) | BOTOX® 72U (N=38) | BOTOX® 48U (N=37) | BOTOX® 24U (N=37) | Placebo (N=37)
Facial paresis (Nervous system disorders) | 4 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 2 | 1 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 0
Injection site pain (General disorders) | 1 | 1 | 2 | 1 | 0
Mastication disorder (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4 | 2 | 1
Influenza (Infections and infestations) | 0 | 3 | 0 | 5 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 7 | 4 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 3 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2014-02-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT02010775/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT02010775/SAP_001.pdf